CLINICAL TRIAL: NCT07102290
Title: Texting to Recruit Unassisted Tobacco Users at a Large Safety Net Health System Into Quitline Service for a Medicaid Value-based Care Program: Pragmatic Randomized Controlled Trial
Brief Title: Pragmatic Trial of Text Messages to Recruit Unassisted Tobacco Users Into Quitline Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Kick It California (Unknown); Los Angeles County Department of Public Health (Other Government); Tobacco Related Disease Research Program (Other); California Smokers' Helpline (Other)
Responsible Party: Principal Investigator, Elisa Tong, MD, Professor, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1301241
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Smoking Cessation Counselling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Free counseling text message (Placebo Comparator): Usual care of free quitline counseling
  Interventions: Behavioral: Free Help
- Free nicotine patch text message (Active Comparator): Medication incentive offer with free quitline counseling
  Interventions: Behavioral: Free Nicotine message
- Spanish Arm: Free counseling text message (Placebo Comparator): Usual care of free quitline counseling
  Interventions: Behavioral: Spanish: Free help message
- Spanish Arm: Free nicotine patch message (Active Comparator): Medication incentive offer with free quitline counseling
  Interventions: Behavioral: Spanish: Free nicotine message

INTERVENTIONS:
Behavioral: Free Help — Text message offering free quitline coaching. FREE HELP: Hello #first name#, Kick It California works with your provider to help you quit smoking at no cost. A Quit Coach can double your chances of quitting. For more info call 1-844-XXXXXXX.
  Arms: Free counseling text message
Behavioral: Free Nicotine message — Text message for free nicotine patches with free quitline counseling. FREE NRT: Hello #first name#, Kick It California works with your provider to help you quit smoking at no cost. You may be able to get nicotine patches mailed to your home at no cost. For more info call 1-844-XXXXXXX.
  Arms: Free nicotine patch text message
Behavioral: Spanish: Free help message — (Spanish translation available as only English text can be published online in clincialtrials.gov): Text message offering free quitline coaching. FREE HELP: Hello #first name#, Kick It California works with your provider to help you quit smoking at no cost. A Quit Coach can double your chances of quitting. For more info call 1-844-XXXXXXX.
  Arms: Spanish Arm: Free counseling text message
Behavioral: Spanish: Free nicotine message — (Spanish translation available as only English text can be published online in clinicaltrials.gov): Text message for free nicotine patches with free quitline counseling. FREE NRT: Hello #first name#, Kick It California works with your provider to help you quit smoking at no cost. You may be able to get nicotine patches mailed to your home at no cost. For more info call 1-844-XXXXXXX.
  Arms: Spanish Arm: Free nicotine patch message

SUMMARY:
The goal of this pragmatic trial is to compare the effects of text messages on quitline enrollment by patients identified in electronic health records as unassisted tobacco users. The main question it aims to answer is:

Do messages offering free counseling or free nicotine patches by text increase quitline enrollment?

Researchers will compare if people receiving texts about free nicotine patches will have higher quitline enrollment than texts about free counseling.

Participants will receive a text message stratified by quitline language and click on the toll-free number to access quitline services.

DETAILED DESCRIPTION:
Participants were patients of Los Angeles County Department of Health Services (LADHS). Through the LADHS population health team, eligible patients were identified through data extraction from the electronic health record for quality metric reporting.

Participants were stratified by language (English, Spanish) by LADHS, then randomly assigned to one of two groups. The randomization assignment was generated by a statistician from Kick It California, and text messages were assigned to groups and delivered by LADHS.

Group 1 received a text message offering free quitline coaching. Group 2 received a text message offering free nicotine patches. The texts were sent April-May 2022 and were in English or Spanish according to patient preference. All messages contained a toll-free number to access services, which could be called directly from the text message link, but for tracking purposes different numbers were used.

The quitline, Kick It California, offered coaching to all enrolled participants. The quitline also mailed a 2-week supply of nicotine patches to all enrolled participants unless contraindicated, regardless of which text offer they received. To ensure equitable access, a second text was sent to all participants in June 2022 offering free NRT.

ELIGIBILITY:
Inclusion Criteria:

* Patient of Los Angeles County Department of Health Services with clinical encounter in past 12 months
* 18 years or older
* English or Spanish language
* Had cell phone
* Permission to text
* Patient identified as tobacco user with no documented assistance (e.g., smoking cessation medication, quitline referral, brief counseling by provider) in the prior 24 months

Exclusion Criteria:

- Languages other than English or Spanish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4171 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Calls to the quitline | 1 month
  Proportion of patients (identified as a tobacco user who has not received cessation assistance) calling the quitline from the link in the text message

SECONDARY OUTCOMES:
Receipt of quitline treatment | 1-3 months
  Proportion of patients (identified as tobacco user who has not received cessation assistance) who called the quitline from a text message and received evidence-based cessation treatments (e.g., quitline coaching, nicotine replacement therapy medication, or both)

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Tong, MD, Principal Investigator — University of California, Davis
Locations (1):
- Kick It California, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data about people who engaged with quitline services may be shared if permitted by the quitline protocol, please contact Kick It California
Supporting Information: Study Protocol, SAP
Time Frame: Start date: 8/1/2025, End date: 7/31/2026
Access Criteria: People interested to access the IPD and supporting information will need to contact the study investigators and Kick It California

REFERENCES:
- See also: Related Info — https://www.kickitca.org